CLINICAL TRIAL: NCT01444638
Title: Evaluation of US Assistance for Anesthesia Trainees for Spinal Placement in Parturients Having Caesarean Section: A Randomized Control Trial
Brief Title: Evaluation of Ultrasound (US) Assistance for Anesthesia Trainees for Caesarean Section Spinal Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Timothy Turkstra, Assistant Professor, Staff Anesthesiologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: R-10-594; 17529 (Other: REB)
Record Dates: First submitted 2011-08-03; First posted 2011-10-03 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Pregnancy
Keywords: pregnancy; Caesarian; section; spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental): Trainees will receive pre-procedure U/S guided examination of the parturient's back.
  Interventions: Device: Ultrasound examination
- Control (No Intervention): Control group. (Standard practice) Trainees will NOT receive pre-procedure U/S guided examination.

INTERVENTIONS:
Device: Ultrasound examination — Trainees will receive pre-procedure U/S guided examination of the parturient's back.
  Other Names: M-turbo
  Arms: Ultrasound

SUMMARY:
Parturients receiving spinal anesthetic for Cesarean section will be randomized to have/not have pre-spinal ultrasound examination of their back.

DETAILED DESCRIPTION:
Parturients receiving spinal anesthetic for elective Cesarean section will be randomized to have/not have pre-spinal ultrasound examination of their back, prior to spinal insertion by anesthesia trainees.

The hypothesis is that ultrasound visualization of the patient spinal spaces will allow junior residents to correctly place the spinal needle with fewer attempts.

The null hypothesis is that there is no difference in the primary outcome (number of attempts). i.e. the investigators hypothesize that the number of attempts is not affected by ultrasound assistance. The control group will undergo spinal anesthesia with manual palpation, the standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Parturient scheduled for elective spinal anesthetic for caesarean section.
2. Resident level PGY1 or PGY2.
3. Resident experience between 2-25 spinal anesthetics.
4. ASA 1-3 scheduled for elective sections

Exclusion Criteria:

1. Parturient BMI > 40.
2. Emergency C-section.
3. Previous spinal surgery or scoliosis.
4. Parturient refusal
5. Resident refusal
6. Multiple gestations

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of attempts at intrathecal needle tip placement during spinal anesthesia. | Day 1

SECONDARY OUTCOMES:
1. Time to place spinal anesthetic (seconds), measured from introducer placement to confirmation of cerebral spinal fluid (CSF). | Day 1
Space used for 1st attempt, as estimated by palpation or U/S | Day 1
Number of spaces used | Day 1
Dural depth (cm) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Turkstra, M. Eng, MD, Principal Investigator — UWO
Locations (1):
- Victoria Hospital, London, Ontario, Canada